CLINICAL TRIAL: NCT00755027
Title: A Randomised Placebo-controlled Trial of Rasagiline in Parkinson Disease Patients With Symptoms of Apathy
Brief Title: Rasagiline and Apathy in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIRHSCSP/07/14; 2007-004400-12
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Apathy; Rasagiline
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rasagiline — rasagiline 1 mg daily, oral use, during 12 weeks
  Other Names: Azilect

SUMMARY:
The purpose of this study is to determine whether rasagiline is effective in the treatment of apathy in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of rasagiline in patients with Parkinson's disease (PD) and apathy. Secondary objectives are 1) to evaluate the affective and cognitive response to rasagiline and their correlates to apathy and 2) to investigate the metabolic and neurophysiologic correlates of the behavioural, cognitive and emotional, aspects of apathy in PD. This will be an exploratory, randomized, double-blind, placebo controlled, parallel-group study. 40 PD patients with apathy and without dementia will be recruited. Rasagiline 1 mg or matching placebo will be administered once daily in conjunction with the subjects' usual oral antiparkinsonian medications for up to 12 weeks. Patients will be evaluated at screening (-7 days) and baseline (0), as well as at weeks 4, 8, and 12. A perfusion SPECT will be performed at baseline and at week 12. The study will be conducted at the Movement Disorders Unit of the Neurology Department at Sant Pau Hospital (Barcelona, Spain).

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD optimally treated for their motor deficits with stable doses of L-Dopa and/or dopamine agonists and showing a non-zero score on the item 4 (motivation/initiative) of the Unified Parkinson's Disease Rating Scale (UPDRS)

Exclusion Criteria:

* Dementia associated to PD according to DSM IV criteria. History of primary psychiatric illness or Axis I diagnoses according to the Structured Clinical Interview for DSM-IV
* Patients complaining of acute mood or cognitive fluctuations in response to dopaminergic medication
* Patients treated with any MAO inhibitor (including Selegiline), fluoxetine and fluvoxamine during the previous month before inclusion. Also will be excluded patients with a neurological disorder other than PD, any unstable systemic disease and pregnant or possibly pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the mean change from baseline to study endpoint (week 12) in apathy scores as measured by the Lille Apathy Rating Scale (LARS)and the Apathy Scale | week 12

SECONDARY OUTCOMES:
Secondary outcome measures will include change from baseline to study endpoint on a range of scales assessing apathy, depression, other neuropsychiatric symptoms, cognition, sleepiness and quality of life | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Kulisevsky, MD,PhD, Principal Investigator — Neurology Service at Hospital de la Santa Creu i Sant Pau, Autonomous University of Barcelona (Barcelona, Spain)
Locations (1):
- Fundacio de Gestio Sanitaria de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain